CLINICAL TRIAL: NCT02066558
Title: Basic Research on Carbon Monoxide's Headache Inducing Characteristics and Effects on the Cerebral Arteries and Blood Flow in a Humane Experimental Headache Model
Brief Title: Carbon Monoxide's Headache Inducing Characteristics and Effects on the Cerebral Arteries and Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Nanna Arngrim, MD, medical doctor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-3-2013-194
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Headache; Migraine
Keywords: Carbon monoxide; Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Carbon Monoxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- carbon monoxide (Active Comparator): Inhalation of carbon monoxide up to a carboxyhemoglobin concentration of 12% and 22%.
  Interventions: Other: Carbon monoxide
- placebo (Placebo Comparator): Atmospheric air
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Carbon monoxide — carbon monoxide, 4.7, Purity 99.997, inhalation of carbon monoxide in a volume corresponding to carboxyhemoglobin 10 and 20%, calculated from baseline Hg and body mass.
  Arms: carbon monoxide
Other: Placebo
  Arms: placebo

SUMMARY:
In this study the investigators will research the hypothesis that the gas carbon monoxide induces headache and increases the blood flow velocity in the middle cerebral artery.

DETAILED DESCRIPTION:
To investigate headache score and accompanying symptoms during and after inhalation of carbon monoxide.

With transcranial Doppler imaging, c-scan and laser speckle the investigators will investigate changes in blood flow velocity of the middle cerebral artery (MCA), diameter of the superficial temporal artery (STA), the radial artery and facial skin perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-50
* 50-100 kg

Exclusion Criteria:

* Tension type headache more than once/month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease
* Smoking
* Primary relatives with current or previous migraine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Headache scores | 12 h
  Comparison between carbon monoxide and placebo (atmospheric air)

SECONDARY OUTCOMES:
Blood flow velocity | 0-180 min after inhalation
  Carbon monoxide induced changes in blood flow velocity in the middle cerebral artery before and after inhalation.
Artery circumference | 0-180 min
  Carbon monoxide induced changes in the superficial temporal artery and the radial artery before and after inhalation.
Facial blood flow | 0-180 min
  Carbon monoxide induced changes in facial blood flow before and after inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Arngrim, MD, Principal Investigator — Danish Headache Center, Glostrup Hospital
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark, Denmark